CLINICAL TRIAL: NCT04340349
Title: Low-dose Hydroxychloroquine and Bromhexine: a Novel Regimen for COVID-19 Prophylaxis in Healthcare Professionals (ELEVATE Trial)
Brief Title: Low-dose Hydroxychloroquine and Bromhexine: a Novel Regimen for COVID-19 Prophylaxis in Healthcare Professionals
Acronym: ELEVATE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Julio Granados Montiel, Principal Investigator, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25/20
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hydroxychloroquine; Antimalarials; Enzyme Inhibitors; Antirheumatic Agents
Keywords: SARS-CoV-2; COVID-19; Hydroxychloroquine; BROMHEXINE
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Bromhexine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: DOUBLE BLINDED
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Hydroxychloroquine plus Bromhexine (Experimental): 200 mg of Hydroxychloroquine daily for 2 months 8 mg of Bromhexine every 8 hrs for 2 months
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Bromhexine 8 MG
- Hydroxychloroquine plus Bromhexine (Placebo Comparator): 200 mg of Hydroxycholoroquine daily for 2 months 8 mg of Bromhexine every 8 hrs for 2 months
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Bromhexine 8 MG

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — A daily low dose of Hydroxychloroquine Sulfate. Increase the endosomal pH and inhibits of ACE2 glycosylation receptor.
  Other Names: Evoquin
Drug: Bromhexine 8 MG — TMPRSS2 blocker
  Other Names: Bisolvon

SUMMARY:
This study will investigate the security and efficacy of a daily low dose of hydroxychloroquine and Bromhexine, in preventing the development of the disease from COVID-19 in Health Care Workers at a National Institute of Health In Mexico City.

DETAILED DESCRIPTION:
This study will combine two drugs (hydroxychloroquine and Bromhexine) to see if hydroxychloroquine is better in combination with Bromhexine in preventing the development of the disease from COVID-19 in Health Care Workers at a National Institute of Health In Mexico City. Hydroxychloroquine will be used in a low dose (200 mg every 24 hrs). Bromhexine will be 8mg every 8 hrs. The study groups will be the following: 1) HCQ 200mg/d + BHH placebo 2) HCQ placebo plus BHH placebo

ELIGIBILITY:
Inclusion criteria

* Health personnel working at INR LGII or INCMNSZ who wish to participate in the study and sign the informed consent.
* Over 18 and under 60 years of age, both genders.
* Contacting with suspected or confirmed SARS-CoV-2 infection.
* Normal electrocardiogram.

Exclusion criteria

* Positive quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) test for SARS-CoV-2 at the time of inclusion.
* Panel of IgG or IgM antibodies positive for SARS-CoV-2 at the time of inclusion.
* Development of respiratory symptoms suspicious of SARS-CoV-2 infection during the first 7 days after treatment is initiated, confirmed by qRT-PCR and IgG or IgM antibodies postiver for SARS-CoV-2.
* History of allergies to any hydroxychloroquine or bromhexine related compound or medication.
* Use of immunosuppressors for any reason.
* History of bone marrow transplant.
* Known glucose-6-phosphate dehydrogenase deficiency.
* Chronic kidney disease or glomerular filtration <20ml/min.
* Use of other drugs with reported pharmacological interactions (i.e., digitalis, flecainide, amiodarone, procainamide, or propafenone).
* History of long QT syndrome.
* Electrocardiogram with QTc>500 msec.
* Pregnant or breastfeeding personnel.
* Epilepsy.
* Known liver disease.
* Personnel who have received the Covid-19 vaccine

Elimination criteria

* Personnel who decide to leave the study for any reason not related to adverse events.
* Personnel with incomplete information on the primary outcome (qRT-PCR for SARS-CoV-2).
* Personnel who are relocated to work in another institution.
* Personnel who do not wish to participate in the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of the expression of mRNA SARS-CoV-2 and presence or absence of antibodies anti-SARS-CoV-2 | Day 60
  Primary endpoint will be the proportion of health personnel infected by SARS-CoV-2 at day 60 after starting treatment, in both groups. The infection will be diagnosed using qRT-PCR for relative expression of the mRNA of SARS-CoV-2 and the measure of IgM and IgG antibodies anti-SARS-CoV-2 after day 7 of treatment using rapid test Cellex qSARS-CoV-2 IgG/IgM

SECONDARY OUTCOMES:
Quantification of the expression of mRNA SARS-CoV-2 and presence or absence of antibodies anti-SARS-CoV-2 | Day 90
  The secondary endpoint will be the proportion of health personnel infected 90 days after starting treatment in both groups. The infection will be diagnosed using qRT-PCR for relative expression of the mRNA of SARS-CoV-2 and the measure of IgM and IgG antibodies anti-SARS-CoV-2 after day 7 of the start of treatment using rapid test Cellex qSARS-CoV-2 IgG/IgM

OTHER OUTCOMES:
Positive SARS-CoV-2 result during the treatment | Day 30 and day 90
  The proportion of health personnel positive for SARS-CoV-2 and result in the need for oxygen use, admission to the intensive care unit (ICU), presence of pneumonia by computer tomography scan (CT), death, severe pneumonia defined by the American Thoracic Association, time from hospitalization to recovery in days.
Adverse events | Day 60
  The proportion of health personnel presenting any of the following during the study period: death, nausea, vomiting, abdominal pain, diarrhea, rash, itchy skin, hair loss, lengthening of the QT interval in the electrocardiogram (>500msec), corneal opacity, cardiac arrhythmias, heart failure or kidney failure (renal clearance <20ml/min). The proportion of the compound of adverse events between the groups will be analyed using RR and ARI for 60 days with their respective 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Julio Granados-Montiel, MD, PhD, Principal Investigator — Instituto Nacional de Rehabilitacion
Locations (1):
- National Institute of Rehabilitation, Luis Guillermo Ibarra Ibarra, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Under Mexican Law, we are not able to provide IPD

REFERENCES:
- [Background] Pal M, Berhanu G, Desalegn C, Kandi V. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2): An Update. Cureus. 2020 Mar 26;12(3):e7423. doi: 10.7759/cureus.7423. PMID 32337143
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Luzzi GA, Peto TE. Adverse effects of antimalarials. An update. Drug Saf. 1993 Apr;8(4):295-311. doi: 10.2165/00002018-199308040-00004. PMID 8481216
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Dutta D, Sharma M, Sharma R. Short-term Hydroxychloroquine in COVID-19 Infection in People With or Without Metabolic Syndrome - Clearing Safety Issues and Good Clinical Practice. Eur Endocrinol. 2020 Oct;16(2):109-112. doi: 10.17925/EE.2020.16.2.109. Epub 2020 Oct 6. PMID 33117441
- [Background] Paiardini M, Muller-Trutwin M. HIV-associated chronic immune activation. Immunol Rev. 2013 Jul;254(1):78-101. doi: 10.1111/imr.12079. PMID 23772616
- [Background] Chang R, Sun WZ. Repositioning chloroquine as antiviral prophylaxis against COVID-19: potential and challenges. Drug Discov Today. 2020 Oct;25(10):1786-1792. doi: 10.1016/j.drudis.2020.06.030. Epub 2020 Jul 3. PMID 32629169
- [Background] Juurlink DN. Safety considerations with chloroquine, hydroxychloroquine and azithromycin in the management of SARS-CoV-2 infection. CMAJ. 2020 Apr 27;192(17):E450-E453. doi: 10.1503/cmaj.200528. Epub 2020 Apr 8. No abstract available. PMID 32269021
- [Background] Zanasi A, Mazzolini M, Kantar A. A reappraisal of the mucoactive activity and clinical efficacy of bromhexine. Multidiscip Respir Med. 2017 Mar 20;12:7. doi: 10.1186/s40248-017-0088-1. eCollection 2017. PMID 28331610
- [Background] Depfenhart M, de Villiers D, Lemperle G, Meyer M, Di Somma S. Potential new treatment strategies for COVID-19: is there a role for bromhexine as add-on therapy? Intern Emerg Med. 2020 Aug;15(5):801-812. doi: 10.1007/s11739-020-02383-3. Epub 2020 May 26. PMID 32458206
- [Background] Ravi N, Cortade DL, Ng E, Wang SX. Diagnostics for SARS-CoV-2 detection: A comprehensive review of the FDA-EUA COVID-19 testing landscape. Biosens Bioelectron. 2020 Oct 1;165:112454. doi: 10.1016/j.bios.2020.112454. Epub 2020 Jul 18. PMID 32729549
- [Result] Lai C, Yu R, Wang M, Xian W, Zhao X, Tang Q, Chen R, Zhou X, Li X, Li Z, Li Z, Deng G, Wang F. Shorter incubation period is associated with severe disease progression in patients with COVID-19. Virulence. 2020 Dec;11(1):1443-1452. doi: 10.1080/21505594.2020.1836894. PMID 33108255
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Li C, Ji F, Wang L, Wang L, Hao J, Dai M, Liu Y, Pan X, Fu J, Li L, Yang G, Yang J, Yan X, Gu B. Asymptomatic and Human-to-Human Transmission of SARS-CoV-2 in a 2-Family Cluster, Xuzhou, China. Emerg Infect Dis. 2020 Jul;26(7):1626-1628. doi: 10.3201/eid2607.200718. Epub 2020 Jun 21. PMID 32228809
- [Result] Xu H, Zhong L, Deng J, Peng J, Dan H, Zeng X, Li T, Chen Q. High expression of ACE2 receptor of 2019-nCoV on the epithelial cells of oral mucosa. Int J Oral Sci. 2020 Feb 24;12(1):8. doi: 10.1038/s41368-020-0074-x. PMID 32094336
- [Result] Levy A, Yagil Y, Bursztyn M, Barkalifa R, Scharf S, Yagil C. ACE2 expression and activity are enhanced during pregnancy. Am J Physiol Regul Integr Comp Physiol. 2008 Dec;295(6):R1953-61. doi: 10.1152/ajpregu.90592.2008. Epub 2008 Oct 22. PMID 18945956
- [Result] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Result] Zhan M, Qin Y, Xue X, Zhu S. Death from Covid-19 of 23 Health Care Workers in China. N Engl J Med. 2020 Jun 4;382(23):2267-2268. doi: 10.1056/NEJMc2005696. Epub 2020 Apr 15. No abstract available. PMID 32294342
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Liu Q, Bi G, Chen G, Guo X, Tu S, Tong X, Xu M, Liu M, Wang B, Jiang H, Wang J, Li H, Wang K, Liu D, Song C. Time-Dependent Distribution of Hydroxychloroquine in Cynomolgus Macaques Using Population Pharmacokinetic Modeling Method. Front Pharmacol. 2021 Jan 14;11:602880. doi: 10.3389/fphar.2020.602880. eCollection 2020. PMID 33519466
- [Result] Wang LF, Lin YS, Huang NC, Yu CY, Tsai WL, Chen JJ, Kubota T, Matsuoka M, Chen SR, Yang CS, Lu RW, Lin YL, Chang TH. Hydroxychloroquine-inhibited dengue virus is associated with host defense machinery. J Interferon Cytokine Res. 2015 Mar;35(3):143-56. doi: 10.1089/jir.2014.0038. Epub 2014 Oct 16. PMID 25321315
- [Result] Helal GK, Gad MA, Abd-Ellah MF, Eid MS. Hydroxychloroquine augments early virological response to pegylated interferon plus ribavirin in genotype-4 chronic hepatitis C patients. J Med Virol. 2016 Dec;88(12):2170-2178. doi: 10.1002/jmv.24575. Epub 2016 May 25. PMID 27183377
- [Result] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Result] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Result] Han H, Ma Q, Li C, Liu R, Zhao L, Wang W, Zhang P, Liu X, Gao G, Liu F, Jiang Y, Cheng X, Zhu C, Xia Y. Profiling serum cytokines in COVID-19 patients reveals IL-6 and IL-10 are disease severity predictors. Emerg Microbes Infect. 2020 Dec;9(1):1123-1130. doi: 10.1080/22221751.2020.1770129. PMID 32475230
- [Result] Chude CI, Amaravadi RK. Targeting Autophagy in Cancer: Update on Clinical Trials and Novel Inhibitors. Int J Mol Sci. 2017 Jun 16;18(6):1279. doi: 10.3390/ijms18061279. PMID 28621712
- [Result] Geleris J, Sun Y, Platt J, Zucker J, Baldwin M, Hripcsak G, Labella A, Manson DK, Kubin C, Barr RG, Sobieszczyk ME, Schluger NW. Observational Study of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Jun 18;382(25):2411-2418. doi: 10.1056/NEJMoa2012410. Epub 2020 May 7. PMID 32379955
- [Result] Zahr N, Urien S, Llopis B, Pourcher V, Paccoud O, Bleibtreu A, Mayaux J, Gandjbakhch E, Hekimian G, Combes A, Benveniste O, Saadoun D, Allenbach Y, Pinna B, Cacoub P, Funck-Brentano C, Salem JE. Pharmacokinetics and pharmacodynamics of hydroxychloroquine in hospitalized patients with COVID-19. Therapie. 2021 Jul-Aug;76(4):285-295. doi: 10.1016/j.therap.2021.01.056. Epub 2021 Jan 28. PMID 33558079
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Mareev VY, Orlova YA, Pavlikova EP, Matskeplishvili ST, Akopyan ZA, Plisyk AG, Seredenina EM, Asratyan DA, Potapenko AV, Malakhov PS, Samokhodskaya LM, Mershina EA, Sinitsyn VE, Bulanova MM, Fuks AA, Mareev YV, Begrambekova YL, Kamalov AA. [Combination therapy at an early stage of the novel coronavirus infection (COVID-19). Case series and design of the clinical trial "BromhexIne and Spironolactone for Coronsmall a, CyrillicvirUs Infection requiring hospiTalization (BISCUIT)"]. Kardiologiia. 2020 Sep 7;60(8):4-15. doi: 10.18087/cardio.2020.8.n1307. Russian. PMID 33155953
- [Derived] Granados-Montiel J, Hazan-Lasri E, Franco-Cendejas R, Chavez-Heres T, Silva-Bermudez P, Aguilar-Gaytan R, Manzano-Leon N, Mendez-Maldonado K, Alvarez-Arce A, Martinez-Portilla RJ. New prophylaxis regimen for SARS-CoV-2 infection in health professionals with low doses of hydroxychloroquine and bromhexine: a randomised, double-blind placebo clinical trial (ELEVATE Trial). BMJ Open. 2021 Aug 3;11(8):e045190. doi: 10.1136/bmjopen-2020-045190. PMID 34344672
- See also: Dashboard Mexico 2021 — https://covid19.who.int/region/amro/country/mx

DOCUMENTS (1):
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04340349/ICF_000.pdf